CLINICAL TRIAL: NCT03908060
Title: Clinical Effectiveness and Safety of Intraoperative Methadone in Patients Undergoing Laparoscopic Hysterectomy: a Prospective, Double-blind, Randomised Controlled Trial
Brief Title: Clinical Effectiveness and Safety of Intraoperative Methadone in Patients Undergoing Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01052019
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone; Morphine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation and study medication will be handled by the hospital pharmacy. All research team members, caregiving clinicians and enrolled patients will be blinded to the study allocation arms and the randomisation list will be concealed until all statistical analyses are made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous single-dose methadone (Experimental): A 10 ml syringe with 2 mg/ml of methadone will be prepared and and study drug will be administered as intravenous bolus dose (0.2 mg/kg) corresponding to 1 ml for every 10 kg of ideal body weight (height (cm) - 105).
  Interventions: Drug: Methadone
- Intravenous single-dose morphine (Active Comparator): A 10 ml syringe with 2 mg/ml of morphine will be prepared and study drug will be administered as intravenous bolus dose (0.2 mg/kg) corresponding to 1 ml for every 10 kg of ideal body weight (height (cm) - 105).
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — One intravenous administration of methadone (0.2 mg/kg ideal body weight)
  Arms: Intravenous single-dose methadone
Drug: Morphine — One intravenous administration of morphine (0.2 mg/kg ideal body weight)
  Arms: Intravenous single-dose morphine

SUMMARY:
The role of a single-dose of intraoperative methadone on postoperative pain and opioid consumption in patients undergoing hysterectomy remains scarcely explored. A prospective double-blind, randomised controlled trial investigating the effect of a single-dose of intraoperative methadone in patients scheduled for same day hysterectomy is therefore conducted.

DETAILED DESCRIPTION:
Background with aim: Hysterectomy is the most common major gynaecological procedure in the world and hysterectomy on benign indications are increasingly being performed as same-day surgery. Therefore, perioperative anaesthesia has moved towards the use of very short-acting opioids with the incitement to speed up extubation and facilitate hospital discharge. However, the potential consequence is that more patients experience pain and discomfort.

Methadone has several desirable pharmacological features, and a single intraoperative dose of the long acting opioid could therefore theoretically expand the analgesic window and reduce postoperative opioid consumption compared to the more conventional use of short-acting opioids. The aim of this study is to investigate the effect of a single-dose of intravenous intraoperative methadone on postoperative opioid consumption, pain and side effects in patients scheduled for hysterectomy for benign indications. Our primary hypothesis is that intravenous perioperative methadone reduces opioid consumption (oral cumulative equivalent dose) by 30% during the first 24 postoperative hours compared to intravenous morphine.

Methods: 126 patients will be included in an investigator-initiated, prospective, randomised, double-blind, controlled trial with two arms: an intervention arm (methadone 0.2 mg/kg ideal body weight) and a control arm (morphine 0.2 mg/kg ideal body weight). The study will be GCP-monitored, and is approved by the Danish Health and Medicines Authority (2018-004351-20) and the Central Denmark Region Committees on Health Research Ethics (1-10-72-365-18).

Hypothesis: The results will probably be applicable to other types of surgery involving visceral pain, and thus the present study has the potential to improve the pain management for a large number of patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled for elective laparoscopic hysterectomy for benign indications

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status IV or V
* prolonged QT-interval assessed by electrocardiogram (> 440 milliseconds)
* Existing treatment with medications prolonging the QT-interval
* Hysterectomy due to malignancy or acute bleeding disorders
* Allergy to study drugs
* Preoperative daily use of opioids
* Severe respiratory insufficiency
* Heart failure
* Acute alcohol intoxication/delirium tremens
* Increased intracranial pressure
* Acute liver disease
* Acute abdominal pain
* Liver insufficiency
* Kidney insufficiency
* Treatment with rifampicin
* Breastfeeding
* Inability to provide informed consent.

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption at 24 hours after extubation (cumulative opioid consumption) | 24 hours
  cumulative opioid consumption in oral morphine equivalents
Opioid consumption at 6 hours after extubation (cumulative opioid consumption) | 6 hours
  cumulative opioid consumption in oral morphine equivalents

SECONDARY OUTCOMES:
Pain intensity (NRS, 0-10) at rest and coughing | 0-48 hours after extubation
  Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst imaginable pain)
Postoperative side effects/ adverse events (nausea and vomiting, sedation, hypoventilation, and hypoxemia) | 0-72 hours after extubation
  Number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Friesgaard, MD, PhD, Principal Investigator — Department of Anaesthesiology and Intensive Care, Horsens Regional Hospital
Locations (1):
- Department of Anaesthesiology and Intensive Care, Horsens Regional Hospital, Horsens, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Shear T, Parikh KN, Patel SS, Gupta DK. Intraoperative Methadone for the Prevention of Postoperative Pain: A Randomized, Double-blinded Clinical Trial in Cardiac Surgical Patients. Anesthesiology. 2015 May;122(5):1112-22. doi: 10.1097/ALN.0000000000000633. PMID 25837528
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Deshur MA, Vender JS, Benson J, Newmark RL. Clinical Effectiveness and Safety of Intraoperative Methadone in Patients Undergoing Posterior Spinal Fusion Surgery: A Randomized, Double-blinded, Controlled Trial. Anesthesiology. 2017 May;126(5):822-833. doi: 10.1097/ALN.0000000000001609. PMID 28418966
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Richlin DM, Reuben SS. Postoperative pain control with methadone following lower abdominal surgery. J Clin Anesth. 1991 Mar-Apr;3(2):112-6. doi: 10.1016/0952-8180(91)90007-a. PMID 2039637
- [Background] Chui PT, Gin T. A double-blind randomised trial comparing postoperative analgesia after perioperative loading doses of methadone or morphine. Anaesth Intensive Care. 1992 Feb;20(1):46-51. doi: 10.1177/0310057X9202000109. PMID 1609941
- [Derived] Friesgaard KD, Brix LD, Kristensen CB, Rian O, Nikolajsen L. Clinical effectiveness and safety of intraoperative methadone in patients undergoing laparoscopic hysterectomy: a randomised, blinded clinical trial. BJA Open. 2023 Aug 5;7:100219. doi: 10.1016/j.bjao.2023.100219. eCollection 2023 Sep. PMID 37638083